CLINICAL TRIAL: NCT02239627
Title: Prospective, Randomized, Double Blinded Comparison of the Analgesic Efficacy of Epidural Clonidine Versus Corticosteroid for Low Back Pain
Brief Title: Epidural Clonidine Versus Corticosteroid for Low Back Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: based on interim anaylsis
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1407358518
Record Dates: First submitted 2014-09-10; First posted 2014-09-15 (Estimated); Results first posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-12

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain | interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Steroid (Active Comparator): Epidural steroid injection
  Interventions: Drug: Epidural steroid
- Clonidine (Experimental): Epidural clonidine injection
  Interventions: Drug: Clonidine

INTERVENTIONS:
Drug: Epidural steroid
  Arms: Steroid
Drug: Clonidine
  Arms: Clonidine

SUMMARY:
Low back pain is a common condition, affecting majority of the adults in the United States at some point in their lives. Fortunately, most resolve, even without treatment. However, some suffer from continued or recurrent pain.

For those suffering from continued or recurrent low back pain, numerous treatment options exist. One such option is an epidural injection, particularly when other non-surgical treatment options have failed. An epidural injection is the placement of a needle into the space around the spinal cord with the aid of a live X-Ray machine, followed by an injection of various medications. Typically, the medication that is injected is a steroid, commonly with the combination of local anesthetic medication. Epidural steroid injections, with or without local anesthetic is part of the established standard of care in the United States for those with continued or recurrent low back pain. The steroid is believed to reduce inflammation and edema of the injured or irritated nerves. However, despite the routine use of epidural steroids, the steroid itself is not without risks or side effects. Though rare, the steroids have been associated with complications including osteoporosis, steroid induced myopathy, cataracts and many others. In order to minimize the side effects associated with epidural steroids, limiting the dose and frequency have been outlined.

Clonidine is another medication, commonly used in numerous clinical settings. U. S. Food and Drug Administration approved the medication for epidural use for cancer pain but studies have shown effectiveness in non-cancer pain was well and is routinely used for various conditions. There is growing evidence on the use of epidural clonidine for treatment of pain, including low back pain.

This research will study and compare the effectiveness, if any, of clonidine compared to steroid in an epidural injection for low back pain.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has clinical diagnosis of low back due to intervertebral disc disease, spinal stenosis or herniated disc
2. Subject has average pain score (VAS) at least 5
3. Subject has persistent pain despite conservative care
4. Subjects has experienced pain for at least 1 month
5. 18 years of age or older when written informed consent is obtained
6. Signed Institutional Review Board (IRB) approved informed consent form

Exclusion Criteria:

1. Allergy to clonidine, dexamethasone, ropivicaine or lidocaine
2. Coagulopathy
3. Active Infection
4. Serious neurologic deficit
5. Subject is pregnant or planning on becoming pregnant during the course of the study
6. Subject is member of a vulnerable population
7. Investigator suspects substance abuse that might confound the study results
8. Subject has unresolved major issues of secondary gain (as determined by the investigator)
9. Subject exhibits major psychiatric morbidity, untreated or refractory to treatment as determined by the investigator
10. Currently diagnosed with cognitive impairment, or exhibits any characteristic, that would limit study candidate's ability to assess pain relief or complete study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- West Virginia University Hospitals, Morgantown, West Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated and the PI has left the institution. The numbers presented are what was initially entered by the research team. From data available, 16 participants were enrolled on the study; no information about those participants could be located. No other data could be located and it cannot be determined which arm the16 participants were enrolled in or if they completed the study.
Groups:
- Steroid: Epidural steroid injection
  Epidural steroid
- Clonidine: Epidural clonidine injection
  Clonidine
Period: Overall Study
Arm/Group | Steroid | Clonidine
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated and the PI has left the institution. No results information is available, all efforts were to made to retrieve results information, but were unsuccessful. No study data is available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Steroid | Clonidine | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Measured on Visual Analog Scale (VAS)
Time Frame: 3 months
Population: as for baseline characteristics
Arm/Group | Steroid | Clonidine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Pain Relief
Time Frame: Day 0, 3 weeks, 3 months
Population: as for baseline characteristics
Arm/Group | Steroid | Clonidine
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Level of Disability (Oswestry Back Scale)
Time Frame: 3 weeks, 3 months
Population: as for baseline characteristics
Arm/Group | Steroid | Clonidine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Adverse Events
Time Frame: Day 0, 3 weeks, 3 months
Population: as for baseline characteristics
Arm/Group | Steroid | Clonidine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The study was terminated and the PI has left the institution. No results information is available, all efforts were to made to retrieve results information, but were unsuccessful. No study data is available.
Arm/Group | Steroid | Clonidine
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes